CLINICAL TRIAL: NCT01857388
Title: Implementing a School-based Mental Health Prevention Program in Ugandan Schools
Brief Title: School-Based Mental Health Program Implementation in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Makerere University (Other)
Responsible Party: Principal Investigator, Keng-Yen Huang, Assistant Professor, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-00362
Record Dates: First submitted 2013-05-09; First posted 2013-05-20 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Teacher Mental Health Knowledge; Teacher Skills in Addressing Child Mental Health Problem
Keywords: school-based program, mental health, implementation
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ParentCorps (Experimental): Teachers from Intervention schools will receive ParentCorps training and support.
  Interventions: Behavioral: ParentCorps
- Wait List Control (No Intervention): Teachers from control schools will not receive training and support in Year 1, but will receive training and support in Year 2.

INTERVENTIONS:
Behavioral: ParentCorps
  Arms: ParentCorps

SUMMARY:
Implementation of an adapted ParentCorps program in Ugandan schools will improve school mental health service resources, teachers' knowledge about child mental health, and teachers' classroom behavioral management and parent involvement skills.

DETAILED DESCRIPTION:
Participating schools are randomly assigned to a 6-month long school-based intervention or to a wait-list control group. The intervention focuses on improving teacher's classroom behavioral management practices, parent engagement, and child mental health knowledge.

Teachers are assessed at the beginning and the end of the study, and again after 6 months of intervention. Teachers' parent engagement, mental health knowledge, and behavioral practices in the classroom are assessed through observations and teacher ratings.

ELIGIBILITY:
Inclusion Criteria:

* Early childhood teachers

Exclusion Criteria:

* Not early childhood teachers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change of School Teacher Behaviors | Outcome will be measured 3 times--before interveniton, after intervention (about 6 month after the baseline assessment), and 6-month post intervention (about 6 months after the 2nd evaluation)
  Teacher classroom behavioral management skills and parent engagement practices will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Keng-Yen Huang, PhD, MPH, Principal Investigator — NYU School of Medicine; Janet Nakigudde, PhD, Principal Investigator — Makerere University
Locations (1):
- Makerere University, Kampala, Uganda